CLINICAL TRIAL: NCT04041648
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Dose of L606 for Inhalation in Healthy Subjects
Brief Title: Single Ascending Dose Study for Evaluation of Safety, Tolerability and Pharmacokinetics of L606
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmosa Biopharm Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: PBI L606_2.0
Record Dates: First submitted 2019-07-23; First posted 2019-08-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- placebo (Placebo Comparator): placebo group
  Interventions: Device: L606 Inhalation System; Other: Placebo Solution
- L606 Liposomal inhalation solution (Experimental): Liposomal inhalation solution
  Interventions: Drug: L606 (Liposomal Treprostinil) Inhalation Solution 51ug; Device: L606 Inhalation System

INTERVENTIONS:
Drug: L606 (Liposomal Treprostinil) Inhalation Solution 51ug — Single ascending dose
  Other Names: Drug: L606 (Liposomal Treprostinil) Inhalation Solution
  Arms: L606 Liposomal inhalation solution
Device: L606 Inhalation System — Single ascending dose
  Other Names: Device: L606 Inhalation Solution
Other: Placebo Solution — Single ascending dose
  Arms: placebo

SUMMARY:
The primary objective of this study is to evaluate the Pharmacokinetics, Safety and Tolerability of L606 (Liposomal Treprostinil) Inhalation Solution in Single Ascending Dose study design in healthy volunteers.

DETAILED DESCRIPTION:
L606 (Liposomal Treprostinil) Inhalation Solution and dedicated inhalation system is developed by Pharmosa Biopharm Inc. intended to improve the inconvenience, as one of the greatest impediments to patient satisfaction to current inhaled treprostinil therapy. Pharmosa's liposomal technology offers sustained release of treprostinil which enable bid treatment instead of conventional qid treatment offered by current inhaled treprostinil therapy for treatment of patients with PAH (WHO Group 1).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, 18 to 50 years of age, inclusive, at Screening.
2. Body mass index between 18.5 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check in as assessed by the Investigator (or designee).
4. Ability of the subject to generate spirometry according to minimum ATS/ERS guidance criteria.
5. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in Section 6.6.
6. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
7. Agree to abstain from consuming alcohol from 72 hours prior to Check-in.
8. Agree to refrain from strenuous exercise from 7 days prior to Check-in.
9. Agree to abstain from consuming foods and beverages containing poppy seeds, grapefruit, or Seville oranges from 7 days prior to Check-in.
10. Agree to abstain from consuming caffeine-containing foods and beverages from 48 hours prior to Check-in.
11. Agree to abstain from consuming carbonated drinks (including sparkling water and soda) from 48 hours prior to Check-in and until end of study.

Exclusion Criteria:

1. Clinically relevant abnormalities identified during Screening, physical examination, 12 lead ECG, or laboratory examinations.
2. Clinically significant history of hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, genitourinary, and/or musculoskeletal disease, glaucoma, psychiatric disorder, or any other chronic disease, whether controlled by medication or not.
3. History of anaphylaxis, significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless deemed not clinically significant by the Investigator (or designee).
4. History of postural hypotension, unexplained syncope, or hypertension.
5. History of asthma, chronic obstructive pulmonary disease (COPD), or reactive airways conditions or findings consistent with asthma or COPD on spirometry testing.
6. Blood pressure <90 mmHg systolic or <50 mmHg diastolic after supine for 5 minutes at Screening or Check in upon repeat testing.
7. Blood pressure >150 mmHg systolic or >90 mmHg diastolic after supine for 5 minutes at Screening or Check in upon repeat testing.
8. Pulse rate >100 bpm after supine for 5 minutes at Screening or Check-in upon repeat testing.
9. Have a pre-existing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs. Cholecystectomy is permitted if done at least 10 days before enrollment.
10. Use tobacco- or nicotine-containing products within 6 months prior to Check-in, or have a history of >1 pack cigarettes daily use over multiple years of smoking.
11. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
12. Have a history of alcohol abuse or a history of or current impairment of organ function reasonably related to alcohol abuse.
13. Have a history of or current evidence of abuse of licit or illicit drugs or a positive urine screen for drugs of abuse.
14. Alcohol consumption of >21 units per week. One unit of alcohol equals 12 oz (360 mL) beer, 1.5 oz (45 mL) liquor, or 5 oz (150 mL) wine.
15. Positive urine drug screen (including alcohol and cotinine) at Screening and/or Check-in.
16. Positive hepatitis panel and/or positive human immunodeficiency virus test at Screening.
17. Participation in a clinical study involving administration of an investigational drug (new chemical entity) within 30 days prior to Check-in.
18. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
19. Use or intend to use any prescription medications/products within 14 days prior to Check-in with the exception of hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives, unless deemed acceptable by the Investigator (or designee).
20. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
21. Use or intend to use any nonprescription medications/products or herbal supplements within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee). Use of nonsteroidal anti inflammatory drugs or aspirin is prohibited within 14 days prior to Check-in.
22. Receipt of blood products within 2 months prior to Check-in.
23. Donation of blood, plasma, and platelets, or the loss of a significant volume of blood (>450 mL) within 6 weeks prior to Screening.
24. Poor peripheral venous access.
25. Have a history of bleeding problems or abnormal bleeding tendencies.
26. Platelet or coagulation factor levels below the lower limit of normal, unless considered not clinically significant by the Investigator.
27. Have previously completed or withdrawn from this study or any other study investigating treprostinil, and have previously received the investigational product.
28. History of any recent infection within 2 weeks of Check-in.
29. In the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
The number of treatment-emergent adverse events for L606 and placebo, including abnormal laboratory events | From Pre-dose to Day 10
  Frequency, severity and seriousness of adverse events (AE) including physical examination, incident of laboratory abnormalities, 12-lead ECG parameter and vital sign assessment

SECONDARY OUTCOMES:
AUC0-2hr | From pre-dose to 24 hours post dose
  area under curve from time zero to 2 hours postdose
AUC0-4hr | From pre-dose to 24 hours post dose
  AUC from time zero to 4 hours postdose
AUC0-8hr | From pre-dose to 24 hours post dose
  area under curve from time zero to 8 hours postdose
AUC0-12hr | From pre-dose to 24 hours post dose
  area under curve from time zero to 12 hours postdose
AUC0-24hr | From pre-dose to 24 hours post dose
  area under curve from time zero to 24 hours postdose
AUC0-tlast | From pre-dose to 24 hours post dose
  AUC from time zero to the time of the last quantifiable concentration
AUC0-∞ | From pre-dose to 24 hours post dose
  area under curve from time zero to infinite
Cmax | From pre-dose to 24 hours post dose
  maximum plasma concentration
tmax | From pre-dose to 24 hours post dose
  time to Maximum Plasma Concentration
t1/2 | From pre-dose to 24 hours post dose
  time to half-life
CL/F | From pre-dose to 24 hours post dose
  apparent total plasma clearance
Vz/F | From pre-dose to 24 hours post dose
  apparent volume of distribution during terminal phase

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Hunt, MD, PhD, Principal Investigator — Pharmosa Biopharm Inc.PPD
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No